CLINICAL TRIAL: NCT03341663
Title: The Diagnostic Value of Acupoint Sensitization Based on Stable Angina Pectoris
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, Director, West China Hospital
Other Study IDs: 201781590955
Record Dates: First submitted 2017-10-26; First posted 2017-11-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Stable Angina Pectoris; Acupoint Sensitization; Correlation Analysis; Diagnostic Value
Keywords: Stable Angina Pectoris; Acupoint sensitization; Correlation analysis; Diagnostic value
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Coronary angiography,Canadian Cardiovascular Society angina pectoris classification for the severity of angina and electronic Von Frey instrument for testing the degree of acupoint sensitization — All the interventions were tested for only once

SUMMARY:
Investigators adopt cross-sectional study design to carry out the exemplary research in the aspects of disease diagnosis.This study is designed to confirm the hypothesis "acupoint sensitization is associated with a severity of angina pectoris, which may contribute to the diagnosis of stable angina pectoris". After the eligible participants recruited in group, the coronary artery lesions will be evaluated through coronary angiography and the Canadian Cardiovascular Society(CCS) angina pectoris classification will also be evaluated at the same time. The degree of acupoint sensitization will be tested by the electronic Von Frey instrument by one professional acupuncturist with total 12 acupoints, including Shenmen,Yinxi, Shaohao,Jiquan,Neiguan, Ximen, Quze, Shanzhong, Juque, Jueyinyu, Xinyu, Duyu. Analysis were conducted to explore relationships between the degree of acupoint sensitization, the degree of coronary artery stenosis and CCS angina pectoris classification. Diagnostic value will be further analyzed in the final step.

ELIGIBILITY:
Inclusion Criteria:

* Patients meet the diagnostic criteria of ACC/AHA angina pectoris of coronary heart disease
* The frequency of angina attacks were greater or equal to twice a week over the previous 3 months
* Patients agree to do coronary angiography examination and sign the informed consent.

Exclusion Criteria:

* People with mental disabilities and intelligent obstacle
* Patients who can't accomplish the detection of acupoint sensitization
* Patients with allergic condition, especially the contrast media
* Patients with acute myocardial infarction, unstable angina, during arrhythmia and serious diseases which can affect the blood supply of myocardial
* Patients with skin or peripheral nerve paresthesia, pain or the detect area of skin ulcerate
* Pregnant or lactating women
* Patients who undergoing other clinical trials

Ages: 35 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the department of cardiology in the West China Hospital of Sichuan University
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
The degree of acupoint sensitization | About 1 hour
  The value will be obtained through the electronic Von Frey instrument
The degree of coronary artery stenosis | About 2 hours
  Data will be obtained through coronary angiography
Canadian Cardiovascular Society angina pectoris classification | About 1 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The West China Hospital of Sichuan university, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT03341663/Prot_001.pdf